CLINICAL TRIAL: NCT02281227
Title: Determination of a Proper Needle Entry Point; Effects of Skin Compression With an Indicator on Radiation Exposure Time of Fluoroscopically Guided Transforaminal Epidural Block in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2014-0721
Record Dates: First submitted 2014-10-23; First posted 2014-11-03 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain Due to Spinal Nerve Compression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- compression group (Active Comparator): skin compression with an indicator for determination of needle entry point
  Interventions: Procedure: skin compression
- non-compression group (Active Comparator): non skin compression with an indicator for determination of needle entry point
  Interventions: Procedure: skin compression

INTERVENTIONS:
Procedure: skin compression — skin compression with an indicator for determination of needle entry point

SUMMARY:
To evaluate the effects of skin compression with an indicator at the needle entry point on radiation exposure time of fluoroscopically guided transforaminal epidural block in obese patients

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ≥ 25 kg/m2 BMI who were scheduled for the transforaminal epidural injection

Exclusion Criteria:

* Local anesthetic allergy, coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2015-10-10 (Actual); Study Completion 2015-10-10 (Actual)

PRIMARY OUTCOMES:
Total radiation exposure time | immediately ≤1 sec after the confirmation of successful epidural injection
  Total radiation exposure time during whole epidural procedure.

SECONDARY OUTCOMES:
The number of the needle readjustments | immediately ≤1 sec after the confirmation of successful epidural injection
  The number of the needle readjustments for successful epidural injection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea